CLINICAL TRIAL: NCT03309553
Title: Hearing Norton Sound: A Community Randomized Trial to Address Childhood Hearing Loss in Rural Alaska
Brief Title: Reducing Childhood Hearing Loss in an Alaska Native Population Through a New School Screening and Referral Process That Utilizes Mobile Health and Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norton Sound Health Corporation (Other)
Collaborators: Duke University (Other); Johns Hopkins University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AD-1602-34571; AD-1602-34751 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2017-09-29; First posted 2017-10-13 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The randomization assignments will be kept confidential within the study team until hearing screening day, when masking the referral process assignment will no longer be possible. All outcome assessors, including audiologists and ear, nose, and throat (ENT) surgeons reading telemedicine consults within the Alaska Native healthcare system and study team members performing medical record abstraction, will be masked to intervention allocation. Study team members who read telemedicine consults as a part of their clinical responsibilities will abstain from reading any study-related consults. The results of the school screen, mHealth screen, and audiometric assessments will also be masked, such that study team members performing the mHealth screen or audiometric assessment will be masked to the other results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current Primary Care Referral Process (Active Comparator): In villages randomized to the current primary care process, families will be notified if their children screen positive in exactly the same method each school had been using previously. This process involves a letter home to the parents, either sent with the child or by mail, requesting that the parent/caregiver bring the child to village health clinic for an evaluation. The list of referred children is also given to the Norton Sound Audiology Department, who reaches out to families to schedule appointments during the next available audiology clinic.
  Interventions: Other: Current Primary Care Referral Process
- Expedited Telemedicine Referral (Experimental): In villages randomized to the expedited telemedicine intervention, parents of children who screen positive will receive a phone call from the school or the clinic on the day of screening notifying them of the day and time of their child's telemedicine consultation appointment. Appointments will be made same-day or next-day, with community health aides (CHAs) who have dedicated time blocked off to perform telemedicine consults. Participating children screening positive will be transported to clinic for their appointment with adult chaperones. Parents are encouraged but not required to attend, except for children grades 2 and younger, for whom parental participation will be required. Nonparticipating children in communities assigned to the expedited telemedicine intervention arm will receive standard referral following the current school primary care referral process.
  Interventions: Other: Telemedicine Referral Process

INTERVENTIONS:
Other: Current Primary Care Referral Process — Children who screen positive for hearing loss will receive the same method each school had been using previously. This process involves a letter home to the parents, either sent with the child or by mail, requesting that the parent/caregiver bring the child to village health clinic for an evaluation.
  Arms: Current Primary Care Referral Process
Other: Telemedicine Referral Process — In villages randomized to the expedited telemedicine intervention, parents of children who screen positive will receive a phone call from the school or the clinic on the day of screening notifying them of the day and time of their child's telemedicine consultation appointment. Appointments will be made same-day or next-day, with community health aides (CHAs) who have dedicated time blocked off to perform telemedicine consults. Participating children screening positive will be transported to clinic for their appointment with adult chaperones. Parents are encouraged but not required to attend, except for children grades 2 and younger, for whom parental participation will be required. Nonparticipating children in communities assigned to the expedited telemedicine intervention arm will receive standard referral following the current school primary care referral process.
  Arms: Expedited Telemedicine Referral

SUMMARY:
Hearing loss is a common health problem in Alaska. Up to 75% of children growing up in Alaskan villages experience frequent ear infections, one of the major treatable causes of hearing loss. Children with even mild hearing loss face many challenges. These children often experience speech and language delays and have trouble in school. Teens with hearing loss are more likely to drop out of school, and are at risk for having difficulty finding jobs as adults. Promptly diagnosing and treating hearing loss is important for preventing these consequences. Alaska mandates school-based hearing screening, but many children with hearing loss are not identified by the current screening protocol, and most who are referred never make it into the healthcare system for diagnosis and treatment.

Alaska has already developed innovative strategies to address hearing loss. A network of village health clinics staffed by community health aides provide local care, and telemedicine has been adopted in over 250 village clinics statewide. Despite being widely available, telemedicine has not yet been used in school hearing screenings to speed up the referral process.

Norton Sound Health Corporation has partnered with Duke and Johns Hopkins Universities to explore whether a new school screening and referral process that incorporates mobile, or mHealth, screening and telemedicine referral will reduce childhood hearing loss disparities in the Norton Sound region. Children from kindergarten through 12th grade in 15 Norton Sound villages will receive the current school screening protocol and the new mHealth screen. Villages will then be randomized to continue the current primary care referral process or to adopt telemedicine referral for school screenings. The investigators hypothesize that the new mHealth screening protocol will identify more children with hearing loss, and telemedicine referral will reduce time to diagnosis. By better identifying hearing loss and speeding up diagnosis and treatment, the investigators expect the burden of childhood hearing loss to drop, hearing-related quality of life to improve, and school performance to improve in villages with telemedicine referral compared to current primary care referral villages. If the study shows these positive effects, mHealth screening and the telemedicine referral process could be implemented in school districts across the state of Alaska to reducing childhood hearing loss disparities statewide.

ELIGIBILITY:
Inclusion Criteria:

* Student of the Bering Strait School District (BSSD) in Alaska
* All school-aged children, from Kindergarten through 12th grade in the school district are eligible to participate
* Parental signed consent to undergo routine hearing screening in the school setting
* Verbal assent from children enrolled in the study

Exclusion Criteria:

* Not a student of the Bering Strait School District
* Parental consent for routine hearing screening not obtained
* Verbal assent not obtained

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1481 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Time to diagnosis | From date of screening to date of ICD-10 ear/hearing diagnosis, measured in days, up to 9 months from date of screening in Year 1 and Year 2
  Comparing time to International Classification of Disease, Tenth Edition (ICD-10) ear/hearing diagnosis from date of screening between intervention and active comparator

SECONDARY OUTCOMES:
Change in prevalence of hearing loss | Annual audiometric assessment at Year 1 and Year 2
  Based on audiometric assessment criteria, compared between intervention and active comparator
Change in hearing-related quality of life | Annual questionnaire assessment at Year 1 and Year 2
  Measured using Hearing Environments and Reflection on Quality of Life (HEAR-QL) questionnaire, compared between intervention and active comparator
Change in school performance | 3 times annually in Year 1 and Year 2
  Measure of math and reading performance using AIMSweb, compared between intervention and active comparator

OTHER OUTCOMES:
Sensitivity and specificity of screening protocols | Cross-sectional comparison of concurrent mHealth screening protocol and current school hearing screening protocol to audiometric assessment, measured once at Year 1, all communities combined
  School and mobile health (mHealth) screening to audiometric assessment, all measured on the same day in Baseline at Year 1 before intervention
Prevalence of hearing loss | Baseline at Year 1 before intervention
  Estimating baseline prevalence of hearing loss in school-aged children using audiometric assessments, all communities combined

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Kleindienst Robler, AuD, PhD, Principal Investigator — Norton Sound Health Corporation; Susan D Emmett, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Norton Sound Health Corporation, Nome, Alaska, United States

REFERENCES:
- [Derived] Jin FQ, Huang O, Kleindienst Robler S, Morton S, Platt A, Egger JR, Emmett SD, Palmeri ML. A Hybrid Deep Learning Approach to Identify Preventable Childhood Hearing Loss. Ear Hear. 2023 Sep-Oct 01;44(5):1262-1270. doi: 10.1097/AUD.0000000000001380. Epub 2023 Jun 15. PMID 37318215
- [Derived] Emmett SD, Platt A, Gallo JJ, Labrique AB, Wang NY, Inglis-Jenson M, Jenson CD, Hofstetter P, Hicks KL, Ross AA, Egger JR, Robler SK. Prevalence of Childhood Hearing Loss in Rural Alaska. Ear Hear. 2023 Sep-Oct 01;44(5):1240-1250. doi: 10.1097/AUD.0000000000001368. Epub 2023 Jun 8. PMID 37287104
- [Derived] Robler SK, Platt A, Jenson CD, Meade Inglis S, Hofstetter P, Ross AA, Wang NY, Labrique A, Gallo JJ, Egger JR, Emmett SD. Changing the Paradigm for School Hearing Screening Globally: Evaluation of Screening Protocols From Two Randomized Trials in Rural Alaska. Ear Hear. 2023 Jul-Aug 01;44(4):877-893. doi: 10.1097/AUD.0000000000001336. Epub 2023 Mar 13. PMID 36907833
- [Derived] Hicks KL, Robler SK, Simmons RA, Ross A, Egger JR, Emmett SD. Hearing-related quality of life in children and adolescents in rural Alaska. Laryngoscope Investig Otolaryngol. 2022 Dec 1;8(1):269-278. doi: 10.1002/lio2.973. eCollection 2023 Feb. PMID 36846414
- [Derived] Hicks KL, Robler SK, Platt A, Morton SN, Egger JR, Emmett SD. Environmental Factors for Hearing Loss and Middle Ear Disease in Alaska Native Children and Adolescents: A Cross-Sectional Analysis from a Cluster Randomized Trial. Ear Hear. 2023 Jan-Feb 01;44(1):2-9. doi: 10.1097/AUD.0000000000001265. Epub 2022 Aug 23. PMID 35998103
- [Derived] Marrone NL, Nieman CL, Coco L. Community-Based Participatory Research and Human-Centered Design Principles to Advance Hearing Health Equity. Ear Hear. 2022 Jul-Aug 01;43(Suppl 1):33S-44S. doi: 10.1097/AUD.0000000000001183. Epub 2020 Jun 13. PMID 35724253
- [Derived] Emmett SD, Platt A, Turner EL, Gallo JJ, Labrique AB, Inglis SM, Jenson CD, Parnell HE, Wang NY, Hicks KL, Egger JR, Halpin PF, Yong M, Ballreich J, Robler SK. Mobile health school screening and telemedicine referral to improve access to specialty care in rural Alaska: a cluster- randomised controlled trial. Lancet Glob Health. 2022 Jul;10(7):e1023-e1033. doi: 10.1016/S2214-109X(22)00184-X. PMID 35714630
- [Derived] Robler SK, Inglis SM, Gallo JJ, Parnell HE, Ivanoff P, Ryan S, Jenson CD, Ross A, Labrique A, Wang NY, Emmett SD. Hearing Norton Sound: community involvement in the design of a mixed methods community randomized trial in 15 Alaska Native communities. Res Involv Engagem. 2020 Nov 3;6(1):67. doi: 10.1186/s40900-020-00235-0. PMID 33292651
- [Derived] Emmett SD, Robler SK, Wang NY, Labrique A, Gallo JJ, Hofstetter P. Hearing Norton Sound: a community randomised trial protocol to address childhood hearing loss in rural Alaska. BMJ Open. 2019 Jan 15;9(1):e023078. doi: 10.1136/bmjopen-2018-023078. PMID 30782695
- [Derived] Emmett SD, Robler SK, Gallo JJ, Wang NY, Labrique A, Hofstetter P. Hearing Norton Sound: mixed methods protocol of a community randomised trial to address childhood hearing loss in rural Alaska. BMJ Open. 2019 Jan 22;9(1):e023081. doi: 10.1136/bmjopen-2018-023081. PMID 30674486